CLINICAL TRIAL: NCT01125501
Title: Protandim and the Metabolic Syndrome: A Preliminary Study to Define Protein Signatures That Change Along With Lowered Oxidative Stress Measured as F2 Isoprostanes or TBARS and Inflammation Measured as hsCRP
Brief Title: Protandim and the Metabolic Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: funding not available
Sponsor: SomaLogic, Inc. (Industry)
Collaborators: LifeVantage (Unknown)
Responsible Party: Robert H. Eckel, MD; Professor of Medicine, Univeristy of Colorado Denver
Organization: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: SomaL-028 (withdrawn)
Record Dates: First submitted 2010-05-17; First posted 2010-05-18 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2010-07

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Protandim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Protandim (Active Comparator): one capsule a day for 30 days of protandim given, followed by a wash out period.
  Interventions: Dietary Supplement: Protandim
- Placebo (Placebo Comparator): one capsule a day for 30 days will be given followed by a washout period.
  Interventions: Dietary Supplement: Protandim

INTERVENTIONS:
Dietary Supplement: Protandim — The product Protandim used in this study have ingredients derived from five botanical sources [Bacopa monniera, Silybum marianum (milk thistle), Withania somnifera (Ashwagandha), Camellia sinensis (green tea), and Curcuma longa (turmeric)].

SUMMARY:
Protandim will decrease markers of oxidative stress/inflammation in subjects with metabolic syndrome and proteomics will identify protein profiles that correlate with markers or/changes in oxidative stress.

DETAILED DESCRIPTION:
Evaluate the effects of Protandim on protein profile changes and markers of inflammation and oxidation in subjects (40-60 years of age) with the Metabolic Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age = 40-60 years of age
* Meets at least 3 of the 5 criteria for the metabolic syndrome (as defined by NCEP/ATP III criteria)

NCEP/ATP III criteria

* Central obesity as measured by waist circumference:

  * Men - Greater than 40 inches
  * Women - Greater than 35 inches
* Fasting blood triglycerides greater than or equal to 150 mg/dL
* Blood HDL cholesterol:

  * Men - Less than 40 mg/dL
  * Women - Less than 50 mg/dL
* Blood pressure greater than or equal to 130/85 mmHg or on anti-hypertensive Rx
* Fasting glucose greater than or equal to 100 but < 125 mg/dL

Exclusion Criteria:

* Women taking hormone replacement therapy for post menopause
* Signs or symptoms of acute coronary syndrome
* History of congestive heart failure (prior myocardial infarction, coronary artery disease including stent placement, coronary artery bypass graft, EBCT calcium score of at least 100, or a positive stress test)
* Serum creatinine > 1.5 mg/dL, AST or ALT > 2 times ULN, HgA1c >6.5%, severely depressed or elevated blood cell lines, triglycerides > 500, TSH outside of normal range, elevated calcium, blood pressure > 160/100, urine protein > 30 ,g/dl.
* Concurrent medical conditions/illnesses in which expected life expectancy is 2 years or less and/or are likely to require frequent hospitalizations and treatment adjustments (e.g., cirrhosis, active malignancy, , or highly active rheumatologic condition, lupus, rheumatoid arthritis or chronic obstructive pulmonary disease and diabetes).
* Participation in any other investigational substance or medical device study within 30 days before this trial and/or participation in such entity during this trial.
* Known pregnancy.
* Supplementation with nutraceuticals or if so one month washout before initiating the study before initiating this trial.
* Taking statins or fibrates to lower cholesterol
* Inability or unwillingness to provide written informed consent

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Measure Decrease in Oxidative Stress markers. | every 30 days for 120 days
  the primary purpose of this trial is a preliminary study to examine the relationship to markers of oxidative stress,in response to Protandim, in Metabolic Syndrome.

SECONDARY OUTCOMES:
Protein signatures | every 30 days for 120 days
  evaluating the effects of Protandim on protein profile changes in patients with metabolic syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Eckel, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States